CLINICAL TRIAL: NCT02284217
Title: A Prospective, Open-Label, Non-Randomized, Comparative Study Designed to Evaluate the Accuracy and Safety of HS-1000 Device, a Non-Invasive Intracranial Pressure (ICP) Monitor, in Patients Undergoing Invasive ICP Monitoring Procedure for Various Clinical Conditions
Brief Title: An Evaluation of Non-invasive ICP Monitoring in Patients Undergoing Invasive ICP Monitoring Via an External Ventricular Drainage (EVD) Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HeadSense Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HS-009
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Presence of High Intracranial Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with invasive ICP monitor (EVD) (Experimental): Hospitalized patients who have already been implanted with an invasive ICP monitor. Eligible patients will be enrolled into the study and HS-1000 headset portion of the device will be placed in their ears.
  Interventions: Device: EVD

INTERVENTIONS:
Device: EVD — ICP monitoring will be done in parallel for both HS-1000 and ICP monitoring via an EVD device (per clinical protocol without any change in the patient's management). HS-1000 ICP monitoring intervals will last from 30 minutes to 6 hours, continuously depending on the patient's clinical condition. Each such interval may occur three times a day or more depending on the clinical condition of the patient.

SUMMARY:
Invasive intracranial pressure (ICP) monitoring is highly effective, but involves risks. HS-1000 measures ICP non-invasively by assessing the acoustic properties of the patient's head. HS-1000 device, a proprietary new non-invasive ICP monitor, is expected to safely and accurately monitor ICP with minimal discomfort to patients, and provide information about normal or elevated ICP levels to the physicians.

The study objective is to compare the accuracy and safety profile of HS-1000, a non-invasive ICP monitor, to invasive ICP monitoring via an external ventricular drain (EVD)

DETAILED DESCRIPTION:
HS-1000 device, a proprietary new non-invasive ICP monitor, is expected to safely and accurately monitor ICP with minimal discomfort to patients, and provide information about normal or elevated ICP levels to the physicians

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women subjects, aged 18 years old and over at screening visit
* Patients undergoing invasive ICP monitoring via an external ventricular drainage (EVD) device for clinical management
* Survival expectancy greater than one week
* Subject or legal authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
* Subject or legal authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

* Subject with ear disease, ear trauma
* Subjects with a bony abnormality (skull defect)
* Subjects with severe head trauma in which the location and/or severity of the skull fracture(s), i.e. frank skull fracture or major joint dislocations may jeopardize HeadSense monitoring procedure
* Subjects with cerebral fluid (CSF) leakage from the ear (CSF Otorrhea)
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* For women of childbearing potential: pregnancy (positive pregnancy test) or breast-feeding
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Post-hoc algorithm processing to compare ICP values (mmHg) of the HS-1000 device and invasive ICP monitor collected in each ICP monitoring cycle | 2 months after last patient \ last visit
Incidence of AEs through 48 hours from end of ICP monitoring with HS-1000 device | 48 hours from end of ICP monitoring
Rate of ear infections/irritations coded and graded using the adapted CTCAE dictionary provided to the site Principal Investigator (PI) | 48 hours from end of ICP monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Olivi, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (5):
  - University of Miami Hospital, Miami, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Metro Health, Cleveland, Ohio
- Germany (2):
  - Erlangen University, Erlangen
  - Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No